CLINICAL TRIAL: NCT00140231
Title: Role of Leptin in the Neuroendocrine and Immune Response to Fasting in Humans
Brief Title: Role of Leptin in the Neuroendocrine and Immune Response to Fasting
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH); Amgen (Industry)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2002P000049; 2M01RR001032-30 (NIH); 5R01DK058785-07 (NIH)
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Fasting
Keywords: leptin; fasting; reproductive; neuroendocrine; immune function; energy deficiency associated with short-term fasting
MeSH Terms: conditions — Fasting | interventions — recombinant methionyl human leptin; metreleptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metreleptin (Active Comparator): r-metHuLeptin self-administered subcutaneously
  Interventions: Drug: r-metHuLeptin; Other: placebo
- Placebo (Placebo Comparator): Placebo, administered in same method as active arm.
  Interventions: Drug: r-metHuLeptin; Other: placebo

INTERVENTIONS:
Drug: r-metHuLeptin — recombinant human leptin
  Other Names: metreleptin
Other: placebo — placebo (no active drug)

SUMMARY:
The purpose of this study will be to determine whether giving leptin (r-metHuLeptin) to a person when he or she is fasting will reverse changes in metabolism, and hormone levels, and immune function associated with fasting, which decreases leptin levels.

DETAILED DESCRIPTION:
Leptin is a hormone secreted by fat cells under normal conditions and acts in the brain to decrease appetite and increase energy use. Leptin levels usually go down with fasting. This study will evaluate the secretion of an investigational agent called leptin in lean and overweight individuals while fasting and investigate the potential role of leptin as a regulator of immune function and mediator of the neuroendocrine response to food deprivation in humans. Data derived from these studies will provide insights into the mechanisms underlying altered hormone levels and immune function in malnutrition and obesity and thus may provide the basis for future therapeutic interventions for obesity.

Comparison: fed state vs. fasting state vs. fasting + leptin state

ELIGIBILITY:
Inclusion Criteria:

* Healthy lean women (with body mass indices [BMI] < 25 kg/m2)
* Overweight otherwise healthy men (with BMI > 27 kg/m2)
* Overweight otherwise healthy women (with BMI > 27 kg/m2).

Exclusion Criteria:

* A history of any illness that may affect the concentrations of the hormones to be studied, e.g. infectious diseases, renal or hepatic failure, type 1 or type 2 diabetes mellitus, cancer or lymphoma, hypogonadism, malabsorption or malnourishment, hypo- or hyperthyroidism, hypercortisolism, alcoholism or drug abuse, anemia, or eating disorder
* On medications known to affect the hormones to be measured (glucocorticoids, anti-seizure medications, and thyroid hormones)
* A known history of anaphylaxis or anaphylactoid-like reactions, or a known hypersensitivity to E. coli derived proteins

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2002-10; Primary Completion 2011-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos S Mantzoros, MD, DSc, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan JL, Heist K, DePaoli AM, Veldhuis JD, Mantzoros CS. The role of falling leptin levels in the neuroendocrine and metabolic adaptation to short-term starvation in healthy men. J Clin Invest. 2003 May;111(9):1409-21. doi: 10.1172/JCI17490. PMID 12727933
- [Derived] Bouzoni E, Perakakis N, Connelly MA, Angelidi AM, Pilitsi E, Farr O, Stefanakis K, Mantzoros CS. PCSK9 and ANGPTL3 levels correlate with hyperlipidemia in HIV-lipoatrophy, are regulated by fasting and are not affected by leptin administered in physiologic or pharmacologic doses. Metabolism. 2022 Sep;134:155265. doi: 10.1016/j.metabol.2022.155265. Epub 2022 Jul 9. PMID 35820631
- [Derived] Chrysafi P, Perakakis N, Farr OM, Stefanakis K, Peradze N, Sala-Vila A, Mantzoros CS. Leptin alters energy intake and fat mass but not energy expenditure in lean subjects. Nat Commun. 2020 Oct 13;11(1):5145. doi: 10.1038/s41467-020-18885-9. PMID 33051459
- [Derived] Foo JP, Aronis KN, Chamberland JP, Mantzoros CS. Lack of Day/Night variation in fibroblast growth factor 21 levels in young healthy men. Int J Obes (Lond). 2015 Jun;39(6):945-8. doi: 10.1038/ijo.2014.215. Epub 2014 Dec 26. PMID 25540981
- [Derived] Foo JP, Aronis KN, Chamberland JP, Paruthi J, Moon HS, Mantzoros CS. Fibroblast growth factor 21 levels in young healthy females display day and night variations and are increased in response to short-term energy deprivation through a leptin-independent pathway. Diabetes Care. 2013 Apr;36(4):935-42. doi: 10.2337/dc12-0497. Epub 2012 Nov 27. PMID 23193213
- [Derived] Moragianni VA, Aronis KN, Chamberland JP, Mantzoros CS. Short-term energy deprivation alters activin a and follistatin but not inhibin B levels of lean healthy women in a leptin-independent manner. J Clin Endocrinol Metab. 2011 Dec;96(12):3750-8. doi: 10.1210/jc.2011-1453. Epub 2011 Sep 14. PMID 21917874
- See also: Click here for more information about the Mantzoros Research Group. — http://www.bidmc.org/Research/Departments/Medicine/Divisions/Endocrinology/Laboratories/MantzorosLab.aspx
- See also: Click here for more information about Beth Israel Deaconess Medical Center. — http://www.bidmc.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Iso Fed, Then Fasting w/ Metreleptin, Then Fasting w/ Placebo: Six young, healthy, and lean women (age, 22.8,; BMI,21.7kg/m2) who were eumenor- rheic were enrolled in a clinical researchcenter- based, randomized, cross-over interventional study involving three separate 5-day-long inpatient admissions (22). Six subjects with a cross-over design, enabling paired comparisons, would provide 80% power to detect a difference of 1.4 SD between different conditionsat the conventional
  a=0.05 level. In thefirst admission, the subjects were studied in the isocaloric fed state, whereas in the following two admissions the subjects were studied in the prolonged fasting state for 72 h and were randomized to receive either placebo or metreleptin at replacement doses. A cross-over to the opposite arm took place in the later admission so that all six subjects received both placebo and metreleptin.
  r-metHuLeptin self-administered subcutaneously
  r-metHuLeptin: recombinant human leptin
- Iso Fed, Then Fasting w/ Placebo, Then Fasting w/ Met: Placebo, administered in same method as active arm.
  placebo: placebo (no active drug)
Period: Fed State 1 Day- day5
Arm/Group | Iso Fed, Then Fasting w/ Metreleptin, Then Fasting w/ Placebo | Iso Fed, Then Fasting w/ Placebo, Then Fasting w/ Met
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Washout 8weeks
Arm/Group | Iso Fed, Then Fasting w/ Metreleptin, Then Fasting w/ Placebo | Iso Fed, Then Fasting w/ Placebo, Then Fasting w/ Met
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: First Fasting State 3 Days With Placebo
Arm/Group | Iso Fed, Then Fasting w/ Metreleptin, Then Fasting w/ Placebo | Iso Fed, Then Fasting w/ Placebo, Then Fasting w/ Met
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Washout 8 Weeks
Arm/Group | Iso Fed, Then Fasting w/ Metreleptin, Then Fasting w/ Placebo | Iso Fed, Then Fasting w/ Placebo, Then Fasting w/ Met
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Fasting State With Leptin and Crossover
Arm/Group | Iso Fed, Then Fasting w/ Metreleptin, Then Fasting w/ Placebo | Iso Fed, Then Fasting w/ Placebo, Then Fasting w/ Met
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Iso Fed, Then Fasting w/ Metreleptin, Then Fasting w/ Placebo: r-metHuLeptin self-administered subcutaneously
  r-metHuLeptin: recombinant human leptin
- Iso Fed, Then Fasting w/ Placebo, Then Fasting w/ Metreleptin: Placebo, administered in same method as active arm.
  placebo: placebo (no active drug)
- Total: Total of all reporting groups
Arm/Group | Iso Fed, Then Fasting w/ Metreleptin, Then Fasting w/ Placebo | Iso Fed, Then Fasting w/ Placebo, Then Fasting w/ Metreleptin | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (5) | 25 (5) | 25.5 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Cortisol
Time Frame: four days
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | Metreleptin | Placebo
Number analyzed (Participants) | 13 | 13
ug/dl | 17.5 (0.9) | 16.9 (1.9)

2. Primary Outcome: ACTH Mean Level
Description: Response of ACTH to leptin administration in fed and fasting state from baseline was measured
Time Frame: 4 days
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Metreleptin | Placebo
Number analyzed (Participants) | 13 | 13
pg/ml
  baseline fed | 10.48 (1.28) | 9.33 (1.23)
  fasting | 9.89 (2.01) | 8.74 (1.75)

3. Primary Outcome: Immune Function CD3 Count
Time Frame: 4 days
Measure: Mean (Standard Error); unit: cells/ul
Arm/Group | Metreleptin | Placebo
Number analyzed (Participants) | 13 | 13
cells/ul | 302 (185) | 838 (268)

4. Secondary Outcome: %Fat Mass
Time Frame: four days
Measure: Mean (Standard Deviation); unit: fat%
Arm/Group | Metreleptin | Placebo
Number analyzed (Participants) | 13 | 13
fat% | 29.1 (2.2) | 29.3 (1.9)

5. Secondary Outcome: (RMR)
Description: Resting Metabolic rate using calorimetry
Time Frame: four days
Measure: Mean (Standard Deviation); unit: kcal/d
Arm/Group | Metreleptin | Placebo
Number analyzed (Participants) | 13 | 13
kcal/d | 1.344 (34) | 1.352 (43)

6. Secondary Outcome: Autonomic Function
Description: aldosterone level were measured on day 4 in response to leptin in fed and fasting states and compared with baseline level on day 1
Time Frame: four days
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Metreleptin | Placebo
Number analyzed (Participants) | 13 | 13
pg/ml
  Day 4 | 132 (27.0) | 112 (23.5)
  day 1 baseline | 66.1 (11.7) | 66.0 (12.8)

ADVERSE EVENTS:
Arm/Group | Metreleptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Our study is confined to lean, healthy female subjects; therefore, our results should not be generalized to male, obese,or diabetic subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No